CLINICAL TRIAL: NCT02242955
Title: Impact of a One-month Long Detoxification Diazepam Treatment on Early Alcohol Relapse
Acronym: DIAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011_44; 2012-003336-23 (EudraCT Number)
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Alcoholism
Keywords: Alcohol-dependence; Relapse; Detoxification; Diazepam; Benzodiazepines; Anxiety
MeSH Terms: conditions — Alcoholism; Recurrence; Anxiety Disorders | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AD = "as-usual diazepam" (Active Comparator): Diazepam treatment duration will not exceed 10 days (commonly recommended duration for alcohol detoxification).
  Interventions: Drug: Diazepam
- PD = "prolonged diazepam" (Experimental): Diazepam will be slowly tapered to be stopped at day 30
  Interventions: Drug: Diazepam

INTERVENTIONS:
Drug: Diazepam — 40 mg per day.

SUMMARY:
Alcohol-dependence is a medical condition that can lead to the occurrence of an alcohol withdrawal syndrome (AWS) in case of alcohol drinking cessation. Diazepam is the reference medication for preventing or treating AWS. The recommended average diazepam treatment duration is usually around one week, and this duration is generally not considered to impact the subsequent relapse rate in alcohol drinking.

However, several previous studies have found that patients experienced frequent anxious symptoms during the weeks following detoxification. Such symptoms may foster early relapse in alcohol drinking. Furthermore, it has been suggested that this anxiety could pertain to late withdrawal symptoms.

The DIAMA study hypothesizes that extending the diazepam detoxification treatment to one month can significantly reduce the cumulated relapse rate in alcohol drinking over the three following months.

DETAILED DESCRIPTION:
* inclusion at Day 5 of the outpatient alcohol detoxification procedure
* randomization in two arms: 1) "10 day - diazepam"; and 2) "30 day - diazepam"
* tapering of diazepam over the 10 days following the beginning of the detoxification procedure in the first arm; tapering of diazepam over the 30 days following the beginning of the detoxification procedure in the second arm.
* 3-month-long follow-up after detoxification. Objective of maintaining abstinence from alcohol. No use of additional anticraving drug. Standardised psychotherapeutic support based on the BRENDA model.
* Longitudinal recording of alcohol consumption using the Alcohol Timeline Follow-Back method.
* Assessment of craving (Obsessive-Compulsive Drinking Scale) and anxiety (State-Trait Anxiety Inventory; Hamilton Anxiety Rating Scale) at Days 5 (baseline), 15, 30, 60 and 90 (final assessment).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-Tr criteria for alcohol dependence
* Diazepam-based outpatient detoxification procedure started 5 days prior to inclusion

Exclusion Criteria:

* contraindication for outpatient detoxification
* occurrence of delirium tremens or seizures during the pre-inclusion period
* contraindication for using diazepam
* any other DSM-IV-TR criteria for substance abuse or dependence in the preceding year (except from tobacco)
* concurrent axis-I psychiatric disorder
* concurrent neurological pathology or cognitive impairment
* concurrent social risk, i.e., homelessness or social isolation
* liver failure, cancer, or significant breathing disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Rate of relapse in alcohol drinking | at 3 months
  Proportion of patients who will have reported any alcohol drinking over the three months following the beginning of the detoxification procedure (using the alcohol timeline follow-back method).

SECONDARY OUTCOMES:
Occurrence of adverse events | Over the first month, at 3 months
Rate of relapse in heavy drinking | at 1 month; at 3 months
  Proportion of patients who will have reported at least one heavy drinking day, i.e., ≥ 50 g of alcohol in a day, over the first month and the three month following the beginning of the detoxification procedure (using the alcohol timeline follow-back method).
Ratio of drinking days/heavy drinking days | over the first month, at 3 months
Level of self-reported anxiety | at 1 month; at 3 months
  Score of self-reported anxiety using the State-Trait Anxiety Inventory
Level of clinician-assessed anxiety | at 1 month; at 3 months
  Score of anxiety using the Hamilton Anxiety Rating Scale
Level of alcohol craving | at 1 month; at 3 months
  Level of alcohol craving using the Obsessive-Compulsive Drinking Scale
Average weekly alcohol consumption | at 1 month; at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, MD, PhD, Principal Investigator — University Hospital of Lille (CHU Lille), France
Locations (2):
- France (2):
  - Department of Addiction Medicine, Lille
  - Outpatient Addiction Center "CSAPA - Le Pari", Lille